CLINICAL TRIAL: NCT04600791
Title: BATwire Implant Kit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Slow enrollment and enough experience gained from the first in human phase of the study and would like to evaluate the findings.
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360058-001
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BATwire Kit (Experimental): Subjects will be implanted using the BATwire Implant Kit
  Interventions: Device: BATwire Implant Kit

INTERVENTIONS:
Device: BATwire Implant Kit — The BATwire Implant Kit is a delivery system for the placement of the Barostim Carotid Sinus Lead.

SUMMARY:
The purpose of this clinical investigation is to develop valid scientific evidence for the safety and effectiveness of the Barostim System delivered by the BATwire Implant Kit (BATwire Kit) in subjects with heart failure. Subjects may be enrolled if they meet the FDA approved PMA indication for use for the Barostim NEO or Barostim NEO2 device: Subjects who remain symptomatic despite treatment with guideline-directed medical therapy, are NYHA Class III or Class II (who had a recent history of Class III), have a left ventricular ejection fraction ≤ 35%, a NT-proBNP < 1600 pg/ml and excludes patients indicated for Cardiac Resynchronization Therapy (CRT) according to AHA/ACC/ESC guidelines.

DETAILED DESCRIPTION:
The BATwire Implant Kit Study is a prospective study of up to 400 subjects enrolled at up to 35 U.S. sites. Up to 100 subjects will be implanted with the Barostim System using the BATwire Kit after all screening is complete and all enrollment criteria are met. The study will evaluate the implant experience, safety and effectiveness of the BATwire kit.

All subjects will be implanted, and the device will be activated prior to being discharged. Follow-up visits will occur at 0.5, 1, 2, 3, 6 and 12 months post implant. Once the 12-month visit has been completed, the subject is withdrawn from the study and followed in a commercial setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 21 years and no more than 80 years at the time of enrollment.
2. Appropriate candidate for the surgery as determined by an evaluation from the implanting physician using a carotid duplex ultrasound (CDU) and/or a computed tomography angiography (CTA), and a review of medical history (including existence of infections that may increase implant risk). Evaluation must confirm the following within 45 days of the Barostim implant (60 days allowed if a proctor is required):

   * Appropriate medical condition and medical history for implantation of the Barostim System AND
   * Anatomy that enables this implant procedure, with no vascular structures or orientations or neck anomalies that would be obstructive to the implantation path AND
   * The artery planned for the Barostim implant must have:

     * A carotid bifurcation below the level of the mandible AND
     * No ulcerative carotid arterial plaques AND
     * No carotid atherosclerosis producing a 30% or greater reduction in linear diameter in the internal carotid AND
     * No carotid atherosclerosis producing a 30% or greater reduction in linear diameter in the distal common carotid AND
   * Have had no prior surgery, radiation, or endovascular stent placement in the carotid artery or the carotid sinus region AND
   * Able to discontinue the use of antiplatelet drugs (e.g., aspirin) in advance of the procedure, if required.
3. Six-minute hall walk (6MHW) ≥ 150 m AND ≤ 400 m within 45 days prior to implant (60 days allowed if a proctor is required).
4. Serum estimated glomerular filtration rate (eGFR) ≥ 25 mL/min/1.73 m^2 using the CKD-EPI method within 45 days prior to the Barostim implant (60 days allowed if a proctor is required).
5. Body mass index ≤ 40 kg/m^2 within 45 days prior to the Barostim implant (60 days allowed if a proctor is required).
6. If female and of childbearing potential, must use a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) and agree to continue use of this method for the duration of the study. Women of childbearing potential must have a negative pregnancy test within 14 days prior to the Barostim implant.
7. Subjects implanted with a cardiac rhythm management device that does not utilize an intracardiac lead, or implanted with a neurostimulation device, must be approved by the CVRx Clinical department.
8. At the end of screening and baseline, the subject still meets the Barostim Indication for Use
9. Signed a CVRx-approved informed consent form for participation in this study.

Exclusion Criteria:

1. Received cardiac resynchronization therapy (CRT) within six months of enrollment, or is actively receiving CRT.
2. Any of the following contraindications:

   * Baroreflex failure or autonomic neuropathy
   * Uncontrolled, symptomatic cardiac bradyarrhythmias
   * Known allergy to silicone or titanium
3. Unstable ventricular arrhythmias.
4. Presence of baseline cranial nerve dysfunction at risk from cervical interventions on the carotid bifurcation determined by the Ear, Nose and Throat (ENT) examination.
5. Subjects with any surgery that has occurred, or is planned to occur, within 45 days of the Barostim implant.
6. Recent history (within 6 months of implant) of significant and uncontrolled bleeding.
7. Known and untreated hypercoagulability state.
8. An inappropriate study candidate as evidenced by:

   * Solid organ or hematologic transplant, or currently being evaluated for an organ transplant.
   * Has received or is receiving LVAD therapy or chronic dialysis.
   * Current or planned treatment with intravenous positive inotrope therapy.
   * Primary pulmonary hypertension.
   * Severe COPD or severe restrictive lung disease (e.g., requires chronic oral steroid use or home oxygen use).
   * Heart failure secondary to a reversible cause, such as cardiac structural valvular disease, acute myocarditis and pericardial constriction.
   * Clinically significant cardiac structural valvular disease.
   * Unable or unwilling to fulfill the protocol medication compliance and follow-up requirements, for reasons including but not limited to an unresolved history of alcohol or substance abuse or psychiatric disorder.
   * Active malignancy.
   * Any other serious medical condition that may adversely affect the safety of the participant or validity of the study, in the opinion of the investigator.
   * Life expectancy less than one year.
9. Any of the following within 3 months prior to the Barostim implant.

   * Myocardial infarction
   * Unstable angina
   * Percutaneous coronary intervention (e.g., CABG or PTCA)
   * Cerebral vascular accident or transient ischemic attack
   * Sudden cardiac death
   * Surgical cardiac intervention (e.g., cardiac ablation, valve replacement)
10. Enrolled and active in another (e.g., device, pharmaceutical, or biological) clinical study unless approved by the CVRx Clinical department.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Freedom from Serious Adverse Events (SAEs) related to the implantation of the lead using the BATwire Implant Kit through 30 days post implant | 30 days post-implant
  To demonstrate the safety of implanting the Barostim lead using the BATwire Implant Kit using all serious adverse events that are related to the BATwire lead implantation that occur between implant, or attempted implant, and 30 days post implant.
Six Minute Hall Walk (6MHW) | 6 months post implant
  To demonstrate that treatment with the Barostim System implanted using the BATwire Implant Kit results in an improvement in 6MHW at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Knight, MD, Study Chair — Northwestern University; Michael Zile, MD, Study Chair — Medical University of South Carolina; Fred Weaver, MD, Study Chair — University of Southern California
Locations (10):
- United States (10):
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - HonorHealth, Scottsdale, Arizona
  - AdventHealth, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Health, Atlanta, Georgia
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Cone Health, Greensboro, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Heart, Austin, Texas

IPD SHARING:
Plan to Share IPD: No